CLINICAL TRIAL: NCT03765268
Title: Neurectomy Vs Nerve Sparing in Open Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Principle investigator, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s9
Record Dates: First submitted 2018-07-13; First posted 2018-12-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Denervation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurectomy (Active Comparator): In this group we did mesh hernioplasty of inguinal hernia with neurectomy of iliohypogastric and ilioinguinal nerve
  Interventions: Procedure: Neurectomy in inguinal hernia repair
- Nerve Sparing (Active Comparator): In this group we did mesh hernioplasty of inguinal hernia with preservation of iliohypogastric and ilioinguinal nerve
  Interventions: Procedure: nerve sparing in inguinal hernia repair

INTERVENTIONS:
Procedure: Neurectomy in inguinal hernia repair — Mesh hernioplasty of inguinal hernia with neurectomy of ilioinguinal and iliohypogastric nerve
  Arms: Neurectomy
Procedure: nerve sparing in inguinal hernia repair — Mesh hernioplasty of inguinal hernia with sparing of ilioinguinal and iliohypogastric nerve
  Arms: Nerve Sparing

SUMMARY:
It is a randomized controlled trial in which we are treating inguinal hernia patients with mesh hernioplasty and either neurectomy of iliohypogastric nerve and ilioinguinal neurectomy or preservation comparing post operative acute or chronic pain

ELIGIBILITY:
Inclusion Criteria:

* patients male, and age between 20 to 70 years Reducible inguinal hernia

Exclusion Criteria:

* Irreducible, obstructed or strangulated hernia uncontrolled diabetes

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
percentage of patients developing chronic inguinodynia | 3 months
  Excruciating Pain measured by visual analog score (with 1 being minimum score and 10 being maximum score) for more than 3 months in inguinal region after open mesh hernioplasty for inguinal hernia

CONTACTS AND LOCATIONS:
Overall Officials: Mahmmood Ayyaz, mbbs, fcps, Study Director — Services Hospital, Lahore
Locations (1):
- Services Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided